CLINICAL TRIAL: NCT02254083
Title: Tolerability and Pharmacokinetics/-Dynamics of 0.5 mg and 1.0 mg (Actual 0.8 mg) of BIBT 986 BS Per Hour Given as IV Infusion Over 32 Hours in Healthy Male Subjects. Placebo Controlled, Double Blind Randomised at Each Dose Level
Brief Title: Tolerability and Pharmacokinetics/-Dynamics of BIBT 986 BS in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1192.2
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (3):
- BIBT 986 BS - low (Experimental)
  Interventions: Drug: BIBT 986 BS - low
- BIBT 986 BS - high (Experimental)
  Interventions: Drug: BIBT 986 BS - high
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBT 986 BS - low
  Arms: BIBT 986 BS - low
Drug: BIBT 986 BS - high
  Arms: BIBT 986 BS - high
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the tolerability of an intravenous infusion of 0.5 and 1.0 mg (actual 0.8 mg) BIBT 986 BS per hour over 32 hours as well as pharmacokinetics and the effect on blood coagulation parameters

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >= 18 and <= 55 years
* BMI >= 18.5 and <= 29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Abnormal PT, TT, aPTT (must be within the normal range after no more than one repeated test), thrombocytes < 150000/μl (two repeats of the first test)
* Evidence of hematuria either macroscopically detectable or microscopic on urinalysis (normal microscopic results after no more than one repeated test)
* Evidence of blood dyscrasia, hemorrhagic diathesis, severe thrombocytopenia, cerebrovascular hemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with hemorrhagic tendencies (e.g. cerebral aneurysm, dissecting aorta, Central nervous system (CNS) trauma, retinopathy, nephrolithiasis)
* Recent or contemplated diagnostic or therapeutic procedures with potential for uncontrollable bleeding (e.g. spinal puncture, lumbar block anaesthesia, surgery of CNS or eye or surgery resulting in large open surfaces) within 14 days before or after drug administration of this clinical trial
* Occult blood in 1 of 3 subsequent faecal samples collected for the pre-study examination
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, within 14 days prior to administration or during the trial
* Participation in another trial with an investigational drug (< 2 months prior to administration or during trial)
* Smoker (> 10 cigarettes or >3 cigars or >3 pipes/day)
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation or loss > 400 mL, < 1 month prior to administration or during the trial
* Excessive physical activities < 5 days prior to administration of study drug or during trial
* Clinically relevant laboratory abnormalities
* Veins unsuited for i.v. puncture and administration of prolonged infusions on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture, etc.)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2003-02; Primary Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 48 hours post dose
CT (concentration of the analyte at the end of drug infusion) | up to 48 hours post dose
Css (steady state concentration of the analyte in plasma following a constant rate infusion) | up to 48 hours post dose
Tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 48 hours post dose
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after single dose administration) | up to 48 hours post dose
t1/2 (Terminal half-life of the analyte in plasma after single dose administration) | up to 48 hours post dose
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable drug plasma concentration after single dose administration) | up to 48 hours post dose
λz (terminal rate constant of the analyte in plasma) | up to 48 hours post dose
MRTinf (mean residence time of the analyte in the body after intravenous infusion) | up to 48 hours post dose
CL (Total clearance of the analyte in plasma following intravascular administration) | up to 48 hours post dose
Vss (Apparent volume of distribution at steady state following intravascular administration) | up to 48 hours post dose
Vz (apparent volume of distribution during the terminal phase λz following intravascular administration) | up to 48 hours post dose
Amount of parent drug eliminated in urine (Ae) | up to 48 hours post dose
Change in activated partial thromboplastin time (aPTT) | up to 48 hours post dose
Change in prothrombin time (PT) | up to 48 hours post dose
Change in ecarin clotting time (ECT) | up to 48 hours post dose
Change in thrombin time (TT) | up to 48 hours post dose
Number of subjects with adverse events | up to 4 days
Number of subjects with clinically significant changes in vital signs | up to 4 days
  Pulse rate, systolic & diastolic blood pressure
Change in International Normalised Ratio (INR) | up to 48 hours post dose
Fraction of administered drug excreted unchanged in urine (fe) | up to 48 hours post dose
CLR (renal clearance of the analyte in plasma following intravascular administration) | up to 48 hours post dose